CLINICAL TRIAL: NCT03684382
Title: Development and Evaluation of a Narrative E-Writing Intervention (NeW-I) for Parents of Children With Chronic Life-Threatening Illness
Brief Title: Narrative E-Writing Intervention (NeW-I) for Parents of Children With Chronic Life-Threatening Illness
Acronym: NeW-I
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanyang Technological University (Other)
Collaborators: KK Women's and Children's Hospital (Other Government); Club Rainbow Singapore (Unknown); Muscular Dystrophy Association Singapore (Unknown); Rare Disorders Society Singapore (Unknown)
Responsible Party: Principal Investigator, Andy Hau Yan Ho, PhD, EdD, Assistant Professor, Nanyang Technological University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB-2018-07-009
Record Dates: First submitted 2018-09-24; First posted 2018-09-25 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Parent of Child With Chronic Life-threatening Illness
Keywords: anticipatory grief intervention; randomized controlled trial; narrative therapy; therapist-facilitated e-counselling

STUDY DESIGN:
Intervention Model Description: Participants who have completed the online consent form, affirmed their study participation and completed the baseline assessments are then randomly allocated to either the NeW-I group or the control group via the online NeW-I platform that is developed for the purpose of this study. Such random assignment reduces the potential of bias.
Masking Description: Consenting participants are randomly allocated to either the intervention or the control group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NeW-I group (Experimental): Participants engage in a weekly structured writing task of 15-30 minutes which provides them an opportunity to reflect on the emotional, practical and financial demands of caregiving, and the means to cope with these challenges (week 1), explore avenues where they can seek information and resources for caregiving (week 2), explore the sources of support which they have within their network of family and friends (week 3) and examine how they (and their children) can rise above illness-related challenges and live their lives as fully as possible (week 4). After participants complete their weekly writing task, the written narrative will be reviewed and edited by the therapist within the next 3-4 days. The revised draft will be shared with the participant along with constructive feedback, empathic support and psychoeducation. In week 5, participants will receive a 'legacy' document and engage in a voice call with the therapist to receive psychosocial support and for closure of therapy.
  Interventions: Other: NeW-I group
- Control group (No Intervention): Participants engage in a weekly unstructured writing task of 15-30 minutes with a single open-ended question for each week which allows them to respond in any manner they find acceptable. Simple empathic weekly feedbacks are provided by the therapist to encourage continuous participation. In week 5, a consolidated document that includes all unedited journal writings together with a brief summary statement of appreciation by the therapist will be given to participants to indicate conclusion of participation.

INTERVENTIONS:
Other: NeW-I group — A 5-week intervention offered to parents of children with chronic life-threatening illness using an internet-based narrative approach with life review elements. After completion of the first four weeks of the intervention, participants will receive a 'legacy' document which is a compiled and edited document of their narrative expression during the first four weeks. This legacy document is structured in a manner that enables participants to find a sense of spiritual well-being and hope in their experience of caring for their child through examination of past experiences and achievements as well as future aspirations.
  Arms: NeW-I group

SUMMARY:
Narrative e-Writing Intervention (NeW-I) is an evidence-based, strength-focused and meaning-oriented approach that aims at enhancing well-being, alleviating burden, and reducing adverse grief outcomes among Singaporean parents caring for a child with chronic life-threatening illness. In collaboration with KK Women's and Children's Hospital and Club Rainbow Singapore, a pilot randomized controlled trial with a built-in qualitative evaluation and feasibility study will be carried out to assess the efficacy of the therapist-facilitated NeW-I protocol and platform among a purposive sample of 66 participants. The findings generated will form the foundation for a full-scale RCT for advancing paediatric palliative care and parental bereavement support.

DETAILED DESCRIPTION:
Background: Conventional grief support interventions for parents whose children are suffering from a chronic life-threatening illness often begin only after the child's death. Despite robust evidence which shows that pre-loss interventions that enhance death preparedness can alleviate psychological distress and prevent adverse grief outcomes among family caregivers of dying patients, there is no known program designed specifically to address the psycho-emotional-spiritual needs of parents facing child loss. And while the National Strategy for Palliative Care in Singapore aims to promote holistic end-of- life care services to patients and their caregivers, vast inadequacy continues to exist in the support provided to parents caring for a dying child in the local context.

Objective and Methods: A novel therapist-facilitated, online intervention is conceived to fill this critical service gap. Adopting an evidence-based approach, the research team has developed a strength-focused and meaning-oriented Narrative e-Writing Intervention (NeW-I) for parents anticipating the death of their child due to a chronic life-threatening condition. The design of NeW-I is informed by an existing body of research (i.e. international systematic review and local qualitative inquiry) that critically examines the lived experience of bereaved parents of children with life- limiting illnesses. NeW-I will be implemented in Singapore in collaboration with KK Women and Child's Hospital and Club Rainbow Singapore. A pilot Randomized Control Trial (RCT) with a built-in accessibility and feasibility study will examine the efficacy of the NeW-I therapeutic protocol for enhancing quality of life, spiritual wellbeing, hope and perceived social support, as well as reducing depressive symptoms, caregiver burden and anticipatory grief among a purposive sample of 66 participants.

Significance: NeW-I aspires to enhance quality of life, spiritual well-being, hope and sense of social support, as well as alleviating depressive symptoms, caregiving burden, and adverse grief outcomes among Singaporean parents facing the terminal illness and eventual death of their sick child. The findings generated will form the foundation of a full-scale RCT for advancing holistic paediatric palliative care and parental bereavement support locally and around the world.

ELIGIBILITY:
Inclusion Criteria:

* Mother or father whose child has been diagnosed with a chronic life-threatening illness between the ages of 0-19 years, with a prognosis of more than 3 months since time of study participation so as to ensure successfully completion of all intervention components before child's death.
* Able to speak, read and write in English, as well as to provide informed consent.

Exclusion Criteria:

* Cannot provide informed consent
* Suffering from severely high levels of depressive symptoms, anxiety and psychological distress (i. e. score of 19 or higher on Patient Health Questionnaire-9 (PHQ-9) or score of 29 or higher on Kessler Psychological Distress Scale (K-10))

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Change in scores on Kemp Quality of Life Scale (KQOL) from baseline | Baseline, immediately after completion of the intervention/control protocol, one month post intervention/control protocol, three months post intervention/control protocol, six months post intervention/control protocol.
  The KQOL is a single-item easily administered, self-rated global measure of quality of life in adults (Siebens et al., 2015)
Change in scores on Functional Assessment of Chronic Illness Therapy-Spiritual Well-Being (FACIT-Sp-12) from baseline | Baseline, immediately after completion of the intervention/control protocol, one month post intervention/control protocol, three months post intervention/control protocol, six months post intervention/control protocol.
  The FACIT-Sp-12 is a 12-item questionnaire that examines the relationships between spiritual well-being, health, and adjustment to chronic illness; it has been successfully used to assess spiritual well-being across a wide range of religious traditions, including those who identify themselves as "spiritual yet not religious" (Bredle, Salsman, Debb, Arnold, & Cella, 2011)
Change in scores on Herth Hope Index (HHI) from baseline | Baseline, immediately after completion of the intervention/control protocol, one month post intervention/control protocol, three months post intervention/control protocol, six months post intervention/control protocol.
  The HHI is a 12-item adapted version of the Herth Hope Scale that is used in clinical settings to assess hope in adults, to assist in the planning and evaluation of effective hope-enhancing strategies (Herth, 1992).
Change in scores on Inventory of Social Support (ISS) from baseline | Baseline, immediately after completion of the intervention/control protocol, one month post intervention/control protocol, three months post intervention/control protocol, six months post intervention/control protocol.
  The ISS is a 5-item self-report questionnaire which assess an individuals's satisfaction with their available social support (Hogan & Schmidt, 2002).
Change in scores on Patient Health Questionnaire-9 (PHQ-9) from baseline | Baseline, immediately after completion of the intervention/control protocol, one month post intervention/control protocol, three months post intervention/control protocol, six months post intervention/control protocol.
  The PHQ-9 is a 9-item self-administered and brief version of the PRIME-MD diagnostic instrument for common mental disorders; it is a reliable and valid clinical and research tool to assess severity of depressive symptoms (Kroenke, Spitzer, & Williams, 2001).
Change in scores on Burden Scale for Family Caregivers-Short Version (BSFC-s) from baseline | Baseline, immediately after completion of the intervention/control protocol, one month post intervention/control protocol, three months post intervention/control protocol, six months post intervention/control protocol.
  The BSFC-s is a 10-item economical instrument for assessing a caregiver's total subjective burden in a short time frame; it is considered an appropriate e outcome measure to evaluate caregiver interventions (Graessel, Berth, Lichte, & Grau, 2014).
Change in scores on Brief Grief Questionnaire (BGQ) from baseline | Baseline, immediately after completion of the intervention/control protocol, one month post intervention/control protocol, three months post intervention/control protocol, six months post intervention/control protocol.
  The BGQ is a 5-item self-report instrument for screening complicated grief in clinical and non-clinical settings; it's validity and reliability has been evaluated on different samples including individuals from Asian countries (Ito et al., 2012; Shear, Jackson, Essock, Donahue, & Felton, 2006).

CONTACTS AND LOCATIONS:
Locations (4):
- Singapore (4):
  - Club Rainbow Singapore, Singapore
  - KK Women's and Children's Hospital, Singapore
  - Muscular Dystrophy Association Singapore, Singapore
  - Rare Disorders Society Singapore, Singapore

REFERENCES:
- [Background] Bredle, J. M., Salsman, J. M., Debb, S. M., Arnold, B. J., & Cella, D. (2011). Spiritual Well-Being as a Component of Health-Related Quality of Life: The Functional Assessment of Chronic Illness Therapy-Spiritual Well-Being Scale (FACIT-Sp). Religions, 2(1), 77-94. https://doi.org/10.3390/rel2010077
- [Background] Dutta O, Tan-Ho G, Choo PY, Ho AHY. Lived experience of a child's chronic illness and death: A qualitative systematic review of the parental bereavement trajectory. Death Stud. 2019;43(9):547-561. doi: 10.1080/07481187.2018.1503621. Epub 2018 Oct 4. PMID 30285557
- [Background] Graessel E, Berth H, Lichte T, Grau H. Subjective caregiver burden: validity of the 10-item short version of the Burden Scale for Family Caregivers BSFC-s. BMC Geriatr. 2014 Feb 20;14:23. doi: 10.1186/1471-2318-14-23. PMID 24555474
- [Background] Herth K. Abbreviated instrument to measure hope: development and psychometric evaluation. J Adv Nurs. 1992 Oct;17(10):1251-9. doi: 10.1111/j.1365-2648.1992.tb01843.x. PMID 1430629
- [Background] Ho, A. H. Y. (2017). A Qualitative Study on the Lived Experience of Bereaved Parents of Young Children with Life Threatening Illness: Advancing Parental Bereavement Support in Singapore and Greater Asia (No. 2017-T1-001-034). Singapore Ministry of Education (MOE) Academic Research Fund (AcRF) Tier 1 Fund.
- [Background] Ho AHY, Car J, Ho MR, Tan-Ho G, Choo PY, Patinadan PV, Chong PH, Ong WY, Fan G, Tan YP, Neimeyer RA, Chochinov HM. A novel Family Dignity Intervention (FDI) for enhancing and informing holistic palliative care in Asia: study protocol for a randomized controlled trial. Trials. 2017 Dec 4;18(1):587. doi: 10.1186/s13063-017-2325-5. PMID 29202863
- [Background] Hogan NS, Schmidt LA. Testing the grief to personal growth model using structural equation modeling. Death Stud. 2002 Oct;26(8):615-34. doi: 10.1080/07481180290088338. PMID 12243195
- [Background] Ito M, Nakajima S, Fujisawa D, Miyashita M, Kim Y, Shear MK, Ghesquiere A, Wall MM. Brief measure for screening complicated grief: reliability and discriminant validity. PLoS One. 2012;7(2):e31209. doi: 10.1371/journal.pone.0031209. Epub 2012 Feb 14. PMID 22348057
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Shear KM, Jackson CT, Essock SM, Donahue SA, Felton CJ. Screening for complicated grief among Project Liberty service recipients 18 months after September 11, 2001. Psychiatr Serv. 2006 Sep;57(9):1291-7. doi: 10.1176/ps.2006.57.9.1291. PMID 16968758
- [Background] Siebens HC, Tsukerman D, Adkins RH, Kahan J, Kemp B. Correlates of a Single-Item Quality-of-Life Measure in People Aging with Disabilities. Am J Phys Med Rehabil. 2015 Dec;94(12):1065-74. doi: 10.1097/PHM.0000000000000298. PMID 25888654
- [Derived] Dutta O, Tan-Ho G, Low XC, Tan THB, Ganapathy S, Car J, Ho RM, Miao CY, Ho AHY. Acceptability and feasibility of a pilot randomized controlled trial of Narrative e-Writing Intervention (NeW-I) for parent-caregivers of children with chronic life-threatening illnesses in Singapore. BMC Palliat Care. 2022 Apr 29;21(1):59. doi: 10.1186/s12904-022-00945-0. PMID 35488270
- [Derived] Ho AHY, Dutta O, Tan-Ho G, Tan THB, Low XC, Ganapathy S, Car J, Ho RM, Miao CY. A Novel Narrative E-Writing Intervention for Parents of Children With Chronic Life-Threatening Illnesses: Protocol for a Pilot, Open-Label Randomized Controlled Trial. JMIR Res Protoc. 2020 Jul 5;9(7):e17561. doi: 10.2196/17561. PMID 32623367